CLINICAL TRIAL: NCT04473339
Title: A Randomized Prospective Trail of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Recurrent Ovarian Cancer Patients With Mutations in Homologous Recombination Repair (HRR) Genes
Brief Title: A Randomized Prospective Trail of HIPEC in Recurrent Ovarian Cancer Patients With HRR Mutation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAI Hongbing (Other)
Responsible Party: Sponsor-Investigator, CAI Hongbing, Dr. Prof., Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020107
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-07

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Ovarian Cancer, Epithelial; Hyperthermic Intraperitoneal Chemotherapy(HIPEC); Homologous Recombination Repair Gene Mutation
Keywords: Homologous Recombination Repair Gene Mutation; hyperthermic intraperitoneal chemotherapy; Epithelial Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRR mt 1 (Experimental): Patients are HRR mutated type, will undergo CRS plus HIPEC and then go on to receive standard platinum-based combination doublet intravenous chemotherapy.
  Interventions: Procedure: CRS+HIPEC
- HRR mt 2 (Experimental): Patients are HRR mutated type, will undergo CRS and then go on to receive standard platinum-based combination doublet intravenous chemotherapy.
  Interventions: Procedure: CRS alone
- HRR wt 3 (Experimental): Patients are HRR wild type, will undergo CRS plus HIPEC and then go on to receive standard platinum-based combination doublet intravenous chemotherapy.
  Interventions: Procedure: CRS+HIPEC
- HRR wt 4 (Experimental): Patients are HRR wild type, will undergo CRS and then go on to receive standard platinum-based combination doublet intravenous chemotherapy.
  Interventions: Procedure: CRS alone

INTERVENTIONS:
Procedure: CRS+HIPEC — Patients will undergo only CRS, HIPEC and IVCT.Patients will receive standard platinum-based combination doublet chemotherapy for 6-8 cycles after CRS and then followed by maintenance therapy.
  A single drug lobaplatin(30mg/m2)will be administered in normal saline via HIPEC and it will be continued for 60 minutes in the hyperthermic phase (41°C-43°C). HIPEC will be performed at the 1st, 3rd and 5th day after CRS. The intravenous chemotherapy(IVCT) will start from 7th-14th day after CRS.
  Arms: HRR mt 1; HRR wt 3
Procedure: CRS alone — Patients will undergo only CRS and IVCT.Patients will receive standard platinum-based combination doublet chemotherapy for 6-8 cycles after CRS and then followed by maintenance therapy.
  Arms: HRR mt 2; HRR wt 4

SUMMARY:
A phase III prospective study with the primary objective to investigate the benefit of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in ovarian cancer patients with mutations in homologous recombination repair (HRR) genes. The target population for this study is patients with recurrent ovarian, peritoneal or fallopian tube cancers undergoing Cytoreductive Surgery (CRS). Patients will be divided into two groups according to HRR genes mutation, each group will be further divided into two sub-groups with different intervention. Patients in Group A are HRR mutated type, sub-group 1 will undergo CRS plus HIPEC and then go on to receive standard platinum-based combination doublet intravenous chemotherapy, sub-group 2 will undergo CRS and then go on to intravenous chemotherapy. Patients in Group B are HRR wild type, sub-group 3 will undergo CRS plus HIPEC and then go on to receive standard platinum-based combination doublet intravenous chemotherapy, sub-group 4 will undergo CRS and then go on to intravenous chemotherapy. All patients will receive maintenance therapy with Niraparib after primary treatment. Prognostic information will be collected for investigation of survival benefits of patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* Karnofsky performance status >50 or World Health Organization performance score < 2
* primary or recurrence ovarian, peritoneal or fallopian tube epithelial cancer; first intra-abdominal recurrence without distant metastasis (including: unique resectable pleural metastasis which are platinum-sensitive; resectable single lymphatic metastasis retroperitoneal or inguinal)
* preoperative platinum-based chemotherapy (carboplatin and paclitaxel, carboplatin and liposomal doxorubicin, gemcitabine, trabectedin or topotecan)
* lesion can be removed completely or residual disease < 0.5 cm
* last chemotherapy finished no more than 12 weeks after surgery
* no hepatic function damage
* white blood cell count ≥3.5*10^9/L; platelet count ≥80*10^9/L; Hemoglobin ≥90g/L
* no contraindication of surgery and anesthesia
* life expectancy ≥ 3 months
* informed consent form signed

Exclusion Criteria:

* age < 18 or >75
* no history of other cancer
* platinum allergy
* distant metastasis
* used anti-angiogenic drug within 8 weeks
* possibility of more than two resection of alimentary canal
* recurrence < 6 months after primary treatment
* histologic type: non epithelial origin
* infection out of control
* follow-up unable to carry on (geographic or psychic)
* cardiac insufficiency or respiratory insufficiency
* has received HIPEC already
* being in other clinical study
* pregnancy or lactation period

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | up to 36 months since diagnosis
  The progression-free survival interval was the time between diagnosis and evidence of recurrent or progressive disease.

SECONDARY OUTCOMES:
Overall Survival | up to 36 months since histological diagnosis
  The overall survival interval was the time between diagnosis and death or last follow-up.
DP9 | the 1 day of histological diagnosis and 9 months after
  The 9 months progression-free survival rate was the rate of no evidence of recurrent or progressive disease at the time of 9 months since histological diagnosis.
DP12 | the 1 day of histological diagnosis and 12 months after
  The 9 months progression-free survival rate was the rate of no evidence of recurrent or progressive disease at the time of 12 months since histological diagnosis.
Serious adverse events, SAEs | surgery and with in 30 days
  Serious adverse events occur within 30 days after surgery, measured with CTCAE 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China